CLINICAL TRIAL: NCT04919577
Title: Predictive Factors for Roux Stasis Syndrome After Distal Gastrectomy With Roux-en-Y Reconstruction in Gastric Cancer Patients: A Retrospective Comparative Cohort
Brief Title: Predictive Factors for Roux Stasis Syndrome
Acronym: PFRSS
Status: Completed | Type: Observational
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Principal Investigator, Wei Fu, Principal, Peking University Third Hospital
Other Study IDs: PekingUTH M2019173
Record Dates: First submitted 2021-05-27; First posted 2021-06-09 (Actual); Last update posted 2021-06-09 (Actual); Status verified 2021-06

CONDITIONS: Gastrostomy
Keywords: Roux stasis syndrome Gastric cancer
MeSH Terms: interventions — X-Rays

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- RSS- Group: Patients without RSS after distal gastrectomy.
  Interventions: Diagnostic Test: X-ray
- RSS+ Group: Patients with RSS after distal gastrectomy.
  Interventions: Diagnostic Test: X-ray

INTERVENTIONS:
Diagnostic Test: X-ray — We defined RSS as (1) the presence of symptoms such as nausea, vomiting, or abdominal fullness, (2) refasting after liquid or semi-liquid diets, (3) imaging methods (X-ray, CT, upper gastroenterography) confirmed without mechanical obstruction. All three conditions must be met at the same time and should occur within 30 days after operation.
  Other Names: CT and Upper Gastroenterography

SUMMARY:
Patients who were pathologically diagnosed with gastric cancer and underwent distal gastrectomy with R-Y reconstruction between March 2014 and March 2021 were retrospectively analyzed. The occurrence of RSS was evaluated and examined for correlations with demographic and clinicopathological data. "R" package was used to build a nomogram.

DETAILED DESCRIPTION:
Patient Selection Ethical approval for this study was obtained from the medical ethics research committee of Peking University Third Hospital (IRB00006761-2019173).

Consecutive patients who were pathologically diagnosed with gastric cancer and underwent distal gastrectomy with R-Y reconstruction between March 2014 and March 2021 at Peking University Third Hospital were retrospectively selected (the detailed screening process was shown in Figure 1).

The exclusion criteria for this study were: (1) patients with distant metastasis, (2) patients with palliative surgery, (3) death occurred within 14 days after operation, (4) patients with primary malignant disease in other organs besides stomach.

Surgical Procedure RY reconstruction was performed after standard distal gastrectomy and D2 lymph node dissection. There are several key steps involved in the RY reconstruction process. Firstly, the jejunum was dissected at 20.2cm (average value) distal to Treitz's ligament. Secondly, a side-to-side antecolic gastrojejunostomy was created using a linear stapler between the gastric stump and the distal segment of jejunum. Finally, an end-to-side or side-to-side jejunostomy was performed in output limb at about 37.2cm (average value) distal to the gastrojejunostomy (Figure 2). A cholecystectomy was performed if the patient had gallbladder-related disease.

Data collection We divided these patients into two group depending on whether RSS occurred and retrospectively analyzed the following items: gender, age, body mass index (BMI), smoking, diabetes, high carcinoembryonic antigen (CEA), hypoproteinemia, hyperlipidemia, operation approach, operation time, cholecystectomy, length of input and output loops, intestinal anastomosis approach, pathological T (pT) stage, lymph node metastasis, pathological stage, lymphovascular invasion, nerve invasion and postoperative hospital stay. According to the standard classification of BMI in China11, we divided patients into three groups, including underweight group (BMI < 18.5 kg/m2), obesity group (BMI ≥ 28.0 kg/m2) and normal group (18.5 kg/m2 ≥ BMI < 28.0 kg/m2). The cancer stage was defined according to the 8th cancer Edition Cancer Staging System presented by American Joint Committee on Cancer.

Identification of RSS We defined RSS as (1) the presence of symptoms such as nausea, vomiting, or abdominal fullness, (2) refasting after liquid or semi-liquid diets, (3) imaging methods (X-ray, CT, upper gastroenterography) confirmed without mechanical obstruction. All three conditions must be met at the same time and should occur within 30 days after operation.

Two gastroenterologists screened each patient one by one according to the RSS definition. The third gastroenterologist discussed the inconsistent patients and jointly confirmed whether the patient had RSS.

Statistical Analysis Statistical analysis was performed using the SPSS Statistics version 26.0 software program (IBM, USA). Qualitative data were compared using the chi-square test or Fisher's exact test. Quantitative data were tested by nonparametric test with Mann-Whitney U test. We choose the variables with P < 0.1 in univariate analysis and the variables that may be related to RSS clinically to be included in multivariate analysis, using Binary logistic regression analysis (Forward Conditional). Box-Tidwell method was used to verify that the continuous independent variable and the dependent variable logit transform value to be linear relationship (p > 0.05). Linear regression was used to verify that there was no multicollinearity between each independent variable (Tolerance > 0.1, VIF < 10). Based on the logistic regression results, a nomogram for predicting RSS occurrence after radical gastrectomy for distal gastrectomy with RY anastomosis was established, and performance was quantified to determine discrimination and calibration. The model was internally validated using the 1,000 bootstrapping method to obtain relatively unbiased estimates. Nomogram was built using the "rms" package in R version 3.5.2.All tests were bilateral, and P < 0.05 was considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* pathologically diagnosed with gastric cancer
* underwent distal gastrectomy with R-Y reconstruction
* the date of admission is between March 2014 and March 2021
* the admission place is Peking University Third Hospital.

Exclusion Criteria:

* patients with distant metastasis
* patients with palliative surgery
* death occurred within 14 days after operation
* patients with primary malignant disease in other organs besides stomach.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Consecutive patients who were pathologically diagnosed with gastric cancer and underwent distal gastrectomy with R-Y reconstruction between March 2014 and March 2021 at Peking University Third Hospital were retrospectively selected
Sampling Method: Non-Probability Sample
Enrollment: 220 (Actual)
Dates: Start 2014-03-01 (Actual); Primary Completion 2021-03-01 (Actual); Study Completion 2021-05-01 (Actual)

PRIMARY OUTCOMES:
Roux stasis syndrome | 2014.03.01 to 2021.03.01
  Yes or No. We defined RSS as (1) the presence of symptoms such as nausea, vomiting, or abdominal fullness, (2) refasting after liquid or semi-liquid diets, (3) imaging methods (X-ray, CT, upper gastroenterography) confirmed without mechanical obstruction. If all three conditions meet at the same time and occur within 30 days after operation, we choose Yes, otherwise, we choose No.

SECONDARY OUTCOMES:
Age | 2014.03.01 to 2021.03.01
  unit: years. Checking the admission record.
body mass index (BMI) | 2014.03.01 to 2021.03.01
  unit: kg/m^2. Checking the admission record, get the information of weight in kilograms and height in meters, weight/height^2 get the BMI.
smoking, diabetes | 2014.03.01 to 2021.03.01
  Yes or No. Checking the admission record for a history of smoking and diabetes.
operation approach | 2014.03.01 to 2021.03.01
  Open or Laparoscopic. Checking the surgery record.
operation time | 2014.03.01 to 2021.03.01
  unit: min. Checking the anesthesia record.
cholecystectomy | 2014.03.01 to 2021.03.01
  Yes or No. Checking the surgery record to determine if cholecystectomy is complicating.
high carcinoembryonic antigen (CEA) | 2014.03.01 to 2021.03.01
  Yes or No. Checking preoperative laboratory values, if CEA < 5.0 ng/ml choose No, if CEA ≥ 5.0 ng/ml, choose Yes.
hypoproteinemia | 2014.03.01 to 2021.03.01
  Yes or No. Checking preoperative laboratory values, if albumin < 30.0 g/l choose Yes, if albumin ≥ 30.0 g/l , choose No.
length of input and output loops | 2014.03.01 to 2021.03.01
  unit: cm. Checking the surgery record.
intestinal anastomosis approach | 2014.03.01 to 2021.03.01
  End-to-side or Side-to-side. Checking the surgery record.
pathological T (pT) stage | 2014.03.01 to 2021.03.01
  I or II or III. Checking the postoperative pathological report. The cancer stage was defined according to the 8th cancer Edition Cancer Staging System presented by American Joint Committee on Cancer.
lymph node metastasis, lymphovascular invasion, nerve invasion. | 2014.03.01 to 2021.03.01
  Yes or NO. Checking the postoperative pathological report.
postoperative hospital stay | 2014.03.01 to 2021.03.01
  unit: days. Checking the surgery and discharge record. The length of postoperative hospital stay is obtained by subtracting the date of discharge from the date of surgery.
Gender | 2014.03.01 to 2021.03.01
  Male or Female. Checking the admission record.

CONTACTS AND LOCATIONS:
Overall Officials: Wei Fu, MD, Principal Investigator — General Surgery Department, Peking University Third Hospital; Xin Zhou, MD, Principal Investigator — eneral Surgery Department, Peking University Third Hospital
Locations (1):
- General Surgery Department, Peking University Third Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided
We may upload our raw data to Mendeley Data after accepted.